CLINICAL TRIAL: NCT01708005
Title: DIetary Supplements, Executive funcTions and Vitamin D (DIET-D): a Double-blind Randomized Controlled Trial
Brief Title: DIetary Supplements, Executive funcTions and Vitamin D (DIET-D)
Acronym: DIET-D
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Nantes University Hospital (Other); NUTRISANTE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012-A00453-40
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Vitamin D; Cholecalciferol; Lecitone®Se-Vitamin D3
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): 80 participants start the oral intake of Lecitone®Se-Vitamin D3 the day after inclusion and during 24 weeks
  Interventions: Drug: Lecitone®Se-Vitamin D3
- Placebo (Placebo Comparator): 80 participants in this arm start the oral intake of placebo the day after inclusion and during 12 weeks.
  Then, they start the oral intake of Lecitone®Se-Vitamin D3 12 weeks after inclusion until the 24th week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lecitone®Se-Vitamin D3 — Lecitone®Se-Vitamin D3 is a dietary supplement combining the active ingredients in Lecitone®Se and 100 IU of vitamin D3. This dietary supplement comes in capsule form.
  Participants take 2 capsules of Lecitone®Se -Vitamin D3 per day. The dose of vitamin D supplementation will not be adjusted except in case of an adverse event such as hypercalcemia. In this case, vitamin D supplementation is stopped and the participant is released prematurely from the study.
  Arms: Intervention
Drug: Placebo — The comparator is represented by placebo capsules of identical appearance (same size, same color and same smell) that Lecitone®Se-Vitamin D3 capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect after 12 weeks of the oral intake of Lecitone®Se + 200UI/day of D3 vitamin with the effect of a placebo on changes in cognitive performance in Trial Making Test score part B (this test evaluate executive functions of mental flexibility) in older adults with Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Current treatments for Alzheimer's disease (AD) are symptomatic and can only temporarily slow down AD without altering its natural evolution. The development of new therapies has primarily focused on preventing the progression of AD. This therapeutic strategy involves being interested in patients with an early stage of AD such as a mild cognitive impairment (MCI). We hypothesized that the combination of Lecitone®Se with 200 IU/day of vitamin D can slow or even improve cognitive decline, particularly executive functions.

The primary objective of this trial is to compare the effect after 12 weeks of the oral intake of Lecitone®Se-Vitamin D3 with the effect of a placebo on changes in performance obtained in the TMT B in the older adults with a MCI.

The secondary objectives of the study are as follows:

* To compare the effect after 12 weeks of the oral intake of Lecitone®Se-Vitamin D3 with the effect of a placebo on changes in executive performance in patients with a MCI.
* To compare the effect after 12 weeks of the oral intake of Lecitone®Se-Vitamin D3 with the effect of a placebo on changes in variability of stride time in patients with a MCI.
* To compare the effect after 24 weeks of the oral intake of Lecitone®Se-Vitamin D3 with the effect of a placebo and a delay phase of supplementation on changes in executive performance in patients with a MCI.
* To compare the effect after 24 weeks of the oral intake of Lecitone®Se-Vitamin D3 with the effect of a placebo and a delay phase of supplementation on changes in variability of stride time in patients with a MCI.
* To determine the compliance and tolerance of the oral intake of Lecitone®Se-Vitamin D3 in patients with a MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Memory complaints
* No dementia (DSM-IV, NINCDS-ADRDA negative)
* No depression (Geriatric Depression score ≤ 5/15)
* Ability to walk a distance of 15 meters unaided
* Diagnosis of MCI
* To have hypovitaminosis D (i.e. serum 25-hydroxyvitamin D [25OHD]concentration ≤ 30ng/mL)
* To have no hypercalcemia (defined as serum calcium concentration ≥ 2,65mmol/L)
* To have given and signed an informed consent to participate in the trial
* To be affiliated to French Social Security

Exclusion Criteria:

* Others cognitive disorders (untreated thyroid dysfunction, chronic ongoing ethylism, history of syphilis, stroke, severe depressive symptomatology (Geriatric Depression score > 5/15), existence of dementia according to DSM-IV and NINCDS-ADRDA criteria at the time of inclusion)
* Vitamin D supplementation during inclusion
* Contraindications to vitamin D
* Unstable medical condition
* Enrollment in another simultaneous clinical trial
* Civil defense measures underway

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change in executive performance | This outcome is assessed at baseline, 12 and 24 weeks after inclusion.
  Executive performance is measured with Trial Making Test part B (TMT B)

SECONDARY OUTCOMES:
Change in other executive scores | This outcome is assessed at baseline, 12 and 24 weeks after inclusion.
  Test parts A and B, Stoop test, Processing Speed Index
Change in posture | This outcome is assessed at baseline, 12 and 24 weeks after inclusion.
  Time Up & Go, Five Time Sit-to-Stand and spatio-temporal analysis of walking
Between-group comparison of compliance to treatment | This outcome is assessed at baseline, 12 and 24 weeks after inclusion.
  This outcome is assessed together with the serum concentrations of 25OHD and calcium
Change in gait | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  Time Up & Go, Five Time Sit-to-Stand and spatio-temporal analysis of walking
Between-group comparison of tolerance | This outcome is assessed at baseline, 12 and 24 weeks after inclusion
  This outcome is assessed with the serum concentrations of 25OHD and calcium

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD,PhD, Principal Investigator — Angers University Hospital
Locations (1):
- University Hospital, Angers, France